CLINICAL TRIAL: NCT05346419
Title: Risedronate With High-dose Vitamin D Resolves Hyperparathyroidism and Hypovitaminosis D But Not Osteoporosis in Mexican Postmenopausal Patients
Brief Title: Antiresorptive Effect of Treatment With Risedronate and Vitamin D in Postmenopausal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional 1o de Octubre (Other)
Collaborators: National Polytechnic Institute, Mexico (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 118.2021
Record Dates: First submitted 2022-04-15; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Postmenopausal Osteoporosis; Hypovitaminosis D; Hyperparathyroidism
Keywords: Postmenopause; Postmenopausal Osteoporosis; Hypovitaminosis D; Hyperparathyroidism; Risedronate; Osteopenia; Bone Mineral Density; Bone resorption
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Vitamin D Deficiency; Hyperparathyroidism; Bone Diseases, Metabolic; Bone Resorption | interventions — Risedronic Acid; Vitamin D; Drugs, Generic

STUDY DESIGN:
Intervention Model Description: 33 participants between 40 and 78 years old with a diagnosis of postmenopausal osteoporosis or osteopenia with associated hyperparathyroidism, hypovitaminosis or both conditions were selected. All participants were treated for 6 months with risedronate 35 mg and vitamin D 2800 IU once a week, with additional daily vitamin D supplementation of 4000 IU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Postmenopausal Osteopenia-osteoporosis patients (Experimental): All participants were treated for 6 months with risedronate 35 mg and vitamin D 2800 IU once a week, with additional daily vitamin D supplementation of 4000 IU.
  Interventions: Drug: Risedronate; Drug: Vitamin D

INTERVENTIONS:
Drug: Risedronate — Participants received risedronate 35 mg once a week for 6 months.
  Other Names: SERALIS®
Drug: Vitamin D — Participants received 2,800 IU of vitamin D once a week, with additional daily supplementation of 4,000 IU of vitamin D
  Other Names: Generic

SUMMARY:
Osteoporosis is defined as a systemic disease of bone mineralization, characterized by a decrease in bone mineral density that causes bone fragility and increases the risk of fractures during menopause. Recently, a high prevalence of hypovitaminosis D has been found worldwide, which could trigger a state of secondary hyperparathyroidism that can worsen the state of postmenopausal patients with osteoporosis. An open-label, clinical trial was conducted in Mexican women with postmenopausal osteopenia-osteoporosis to determine the efficacy of the combined treatment with risedronate and high-dose vitamin D in improving bone mineral density, hyperparathyroidism, and hypovitaminosis D.

DETAILED DESCRIPTION:
Participants were selected from the climacteric clinic of the regional hospital "1ro de Octubre-Instituto de Seguridad y Servicios Sociales para Los Trabajadores del Estado (ISSSTE)", Mexico. All participants voluntarily accepted to be part of the study and provided written informed consent.This study was approved by the institutional ethical committee of the hospital with registration number COFEPRIS 17 CI 09005135 with the internal registration number 118.2021. Every participant was clinically examined. Their metabolic state was assessed by considering height, weight, body mass index (BMI) and the percentage of Hb1Ac.

33 patients were included among 40 to 78 years with the diagnosis of postmenopausal osteoporosis with associated hyperparathyroidism, hypovitaminosis D or both conditions. All the patients were treated for 6 months with 35 mg of risedronate and 2800 IU of vitamin D once a week, with additional daily supplementation of 4000 IU of vitamin D.

Statical analysis was performed using PAST 3.0 and GraphPad Prism 8.4.3. software. Some statical parameters, such as arithmetic median (µ), and standard deviation (S.D.) were calculated using Excel-Word. Graphics were constructed with GraphPad Prism 8.4.3 and tables were done in Excel-Word. The assigned α value for this study was <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of postmenopausal osteoporosis or osteopenia.
* Participants with a diagnosis of hyperparathyroidism or hypovitaminosis D.
* Participants who accepted to participate and that provided informed consent.

Exclusion Criteria:

* Participants with oncological pathologies.
* Participants with recent fractures.
* Participants with gastric intolerance or hypersensitivity to the drugs.
* Participants were under treatment with another antiresorptive or bone-forming drug, or if they were receiving treatment with thiazide diuretics, lithium, teriparatide or glucocorticoids.
* Participants with Addison's disease, pheochromocytoma or depressive disorders.

Ages: 40 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Remission of hyperparathyroidism | 6 months
  Remission of hyperparathyroidism was considered when serum parathyroid hormone [PTH] values were below 45 pg/mL.
Remission of hypovitaminosis D | 6 months
  Remission of hypovitaminosis D was considered when serum 25-hydroxy vitamin D [25(OH)D] was above 29 pg/ml.
Remission of osteopenia | 6 months
  Osteopenia remission was considered when densitometry T-score values were below -1.
Remission of Osteoporosis | 6 months
  Osteoporosis remission was considered when densitometry T-score values were below -2.4.

SECONDARY OUTCOMES:
Change from baseline serum calcium at 6 months | 6 months
  Calcium was evaluated as a bone mineralization marker.
Change from baseline serum phosphorus at 6 months | 6 months
  Phosphorus was evaluated as a bone mineralization marker.
Change from baseline urinary calcium at 6 months | 6 months
  Urinary calcium was evaluated as an indirect marker of bone demineralization.
Change from bone resorption biomarker at 6 months | 6 months
  Alkaline Phosphatase was evaluated as a bone resorption biomarker.
Fracture Risk Assessment Tool (FRAX®) for hip fracture | 6 months
  Fracture Risk Assessment Tool (FRAX®) for hip fracture was used to determine the 10-year probability of hip fracture. When the predicted risk was greater than 3% was considered a high risk for hip fracture, and when it was lower than 3%, it was considered a low risk for hip fracture.
Fracture Risk Assessment Tool for major osteoporotic fracture (FRAX® Mo) | 6 months
  Fracture Risk Assessment Tool for major osteoporotic fracture (FRAX® Mo) was used to determine the 10-year probability of major osteoporotic fracture (clinical spine, forearm, hip or shoulder fracture). When the predicted risk was greater than 20% was considered a high risk for major osteoporotic fracture, and when it was lower than 20%, it was considered a low risk of major osteoporotic fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Ocampo Godínez, M.D., Ph.D., Study Director — Tissue Bioengineering Laboratory, National Autonomous University of Mexico [UNAM]; Patricia Loranca-Moreno, M.D., M.Sc., Study Director — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE.; Merle Y Hernández-Castañón, M.D., Principal Investigator — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE
Locations (1):
- Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cossio-Bolanos M, Vidal-Espinoza R, Fuentes-Lopez J, Castelli Correia de Campos LF, Andruske CL, Urra-Albornoz C, Alvear Vasquez F, Gomez-Campos R. Reference values for bone density and bone mineral content from 5 to 80 years old in a province of Chile. PeerJ. 2022 Mar 23;10:e13092. doi: 10.7717/peerj.13092. eCollection 2022. PMID 35345584
- [Background] Kanis JA, Cooper C, Rizzoli R, Reginster JY; Scientific Advisory Board of the European Society for Clinical and Economic Aspects of Osteoporosis (ESCEO) and the Committees of Scientific Advisors and National Societies of the International Osteoporosis Foundation (IOF). European guidance for the diagnosis and management of osteoporosis in postmenopausal women. Osteoporos Int. 2019 Jan;30(1):3-44. doi: 10.1007/s00198-018-4704-5. Epub 2018 Oct 15. PMID 30324412
- [Background] Deng W, Han JC, Chen L, Qi WL. Estrogen receptor alpha gene PvuII polymorphism and risk of fracture in postmenopausal women: a meta-analysis. Genet Mol Res. 2015 Feb 13;14(1):1293-300. doi: 10.4238/2015.February.13.8. PMID 25730068
- [Background] Aziziyeh R, Amin M, Habib M, Perlaza JG, McTavish RK, Ludke A, Fernandes S, Sripada K, Cameron C. A scorecard for osteoporosis in four Latin American countries: Brazil, Mexico, Colombia, and Argentina. Arch Osteoporos. 2019 Jun 27;14(1):69. doi: 10.1007/s11657-019-0622-1. PMID 31250192
- [Background] Moschonis G, van den Heuvel EG, Mavrogianni C, Manios Y. Effect of Vitamin D-Enriched Gouda-Type Cheese Consumption on Biochemical Markers of Bone Metabolism in Postmenopausal Women in Greece. Nutrients. 2021 Aug 27;13(9):2985. doi: 10.3390/nu13092985. PMID 34578863
- [Background] Bouloukaki I, Markakis M, Pateli R, Lyronis I, Schiza S, Tsiligianni I. Vitamin D levels in primary care patients: correlations with clinical, seasonal, and quality-of-life parameters. Fam Pract. 2022 Jul 19;39(4):678-684. doi: 10.1093/fampra/cmac012. PMID 35325110
- [Background] Dixit V, Tripathi RL, Dhanwal DK. Lack of secondary hyperparathyroidism in sub-group of vitamin D deficient postmenopausal women: Is VDR gene polymorphism behind this mystery? Diabetes Metab Syndr. 2022 Jan;16(1):102381. doi: 10.1016/j.dsx.2021.102381. Epub 2021 Dec 28. PMID 34995987
- [Background] Lips P, Hosking D, Lippuner K, Norquist JM, Wehren L, Maalouf G, Ragi-Eis S, Chandler J. The prevalence of vitamin D inadequacy amongst women with osteoporosis: an international epidemiological investigation. J Intern Med. 2006 Sep;260(3):245-54. doi: 10.1111/j.1365-2796.2006.01685.x. PMID 16918822
- [Background] Martinez-Zavala N, Lopez-Sanchez GN, Vergara-Lopez A, Chavez-Tapia NC, Uribe M, Nuno-Lambarri N. Vitamin D deficiency in Mexicans have a high prevalence: a cross-sectional analysis of the patients from the Centro Medico Nacional 20 de Noviembre. Arch Osteoporos. 2020 Jun 16;15(1):88. doi: 10.1007/s11657-020-00765-w. PMID 32542548
- [Background] Wihlborg A, Bergstrom K, Gerdhem P, Bergstrom I. Parathyroid Hormone Disturbances in Postmenopausal Women with Distal Forearm Fracture. World J Surg. 2022 Jan;46(1):128-135. doi: 10.1007/s00268-021-06331-w. Epub 2021 Oct 13. PMID 34647149
- [Background] Yalla N, Bobba G, Guo G, Stankiewicz A, Ostlund R. Parathyroid hormone reference ranges in healthy individuals classified by vitamin D status. J Endocrinol Invest. 2019 Nov;42(11):1353-1360. doi: 10.1007/s40618-019-01075-w. Epub 2019 Jul 4. PMID 31273631
- [Background] Clark P, Vivanco-Munoz N, Pina JT, Rivas-Ruiz R, Huitron G, Chico-Barba G, Reza-Albarran AA. High prevalence of hypovitaminosis D in Mexicans aged 14 years and older and its correlation with parathyroid hormone. Arch Osteoporos. 2015;10:225. doi: 10.1007/s11657-015-0225-4. Epub 2015 Jul 14. PMID 26168767
- [Background] Yuan F, Peng W, Yang C, Zheng J. Teriparatide versus bisphosphonates for treatment of postmenopausal osteoporosis: A meta-analysis. Int J Surg. 2019 Jun;66:1-11. doi: 10.1016/j.ijsu.2019.03.004. Epub 2019 Mar 16. PMID 30890377
- [Background] Miller PD, Hattersley G, Riis BJ, Williams GC, Lau E, Russo LA, Alexandersen P, Zerbini CA, Hu MY, Harris AG, Fitzpatrick LA, Cosman F, Christiansen C; ACTIVE Study Investigators. Effect of Abaloparatide vs Placebo on New Vertebral Fractures in Postmenopausal Women With Osteoporosis: A Randomized Clinical Trial. JAMA. 2016 Aug 16;316(7):722-33. doi: 10.1001/jama.2016.11136. PMID 27533157
- [Background] Soreskog E, Lindberg I, Kanis JA, Akesson KE, Willems D, Lorentzon M, Strom O, Berling P, Borgstrom F. Cost-effectiveness of romosozumab for the treatment of postmenopausal women with severe osteoporosis at high risk of fracture in Sweden. Osteoporos Int. 2021 Mar;32(3):585-594. doi: 10.1007/s00198-020-05780-8. Epub 2021 Jan 6. PMID 33409591
- [Background] Miyoshi A, Kameda H, Nagai S, Nakamura A, Miya A, Takase T, Atsumi T, Miyoshi H. Beneficial effects of switching to denosumab from bisphosphonates or selective estrogen receptor modulators in postmenopausal women with type 2 diabetes and osteopenia/osteoporosis. J Diabetes Investig. 2021 Jul;12(7):1293-1300. doi: 10.1111/jdi.13458. Epub 2020 Dec 13. PMID 33141482
- [Background] Eastell R, Rosen CJ, Black DM, Cheung AM, Murad MH, Shoback D. Pharmacological Management of Osteoporosis in Postmenopausal Women: An Endocrine Society* Clinical Practice Guideline. J Clin Endocrinol Metab. 2019 May 1;104(5):1595-1622. doi: 10.1210/jc.2019-00221. PMID 30907953
- [Background] Kobayakawa T, Miyazaki A, Saito M, Suzuki T, Takahashi J, Nakamura Y. Denosumab versus romosozumab for postmenopausal osteoporosis treatment. Sci Rep. 2021 Jun 3;11(1):11801. doi: 10.1038/s41598-021-91248-6. PMID 34083636
- [Background] Hiligsmann M, Reginster JY. Cost-effectiveness of gastro-resistant risedronate tablets for the treatment of postmenopausal women with osteoporosis in France. Osteoporos Int. 2019 Mar;30(3):649-658. doi: 10.1007/s00198-018-04821-7. Epub 2019 Jan 30. PMID 30701342
- [Background] McClung MR, Ebetino FH. History of risedronate. Bone. 2020 Aug;137:115407. doi: 10.1016/j.bone.2020.115407. Epub 2020 May 6. PMID 32387834
- [Background] American Geriatrics Society Workgroup on Vitamin D Supplementation for Older Adults. Recommendations abstracted from the American Geriatrics Society Consensus Statement on vitamin D for Prevention of Falls and Their Consequences. J Am Geriatr Soc. 2014 Jan;62(1):147-52. doi: 10.1111/jgs.12631. Epub 2013 Dec 18. PMID 24350602
- [Background] Jilka RL, Weinstein RS, Bellido T, Roberson P, Parfitt AM, Manolagas SC. Increased bone formation by prevention of osteoblast apoptosis with parathyroid hormone. J Clin Invest. 1999 Aug;104(4):439-46. doi: 10.1172/JCI6610. PMID 10449436
- [Background] Balani DH, Ono N, Kronenberg HM. Parathyroid hormone regulates fates of murine osteoblast precursors in vivo. J Clin Invest. 2017 Sep 1;127(9):3327-3338. doi: 10.1172/JCI91699. Epub 2017 Jul 31. PMID 28758904
- [Background] Brent MB, Stoltenborg FE, Bruel A, Thomsen JS. Teriparatide and Abaloparatide Have a Similar Effect on Bone in Mice. Front Endocrinol (Lausanne). 2021 Apr 19;12:628994. doi: 10.3389/fendo.2021.628994. eCollection 2021. PMID 33953694
- [Background] McClung MR, Harvey NC, Fitzpatrick LA, Miller PD, Hattersley G, Wang Y, Cosman F. Effects of abaloparatide on bone mineral density and risk of fracture in postmenopausal women aged 80 years or older with osteoporosis. Menopause. 2018 Jul;25(7):767-771. doi: 10.1097/GME.0000000000001080. PMID 29462094
- [Background] Neer RM, Arnaud CD, Zanchetta JR, Prince R, Gaich GA, Reginster JY, Hodsman AB, Eriksen EF, Ish-Shalom S, Genant HK, Wang O, Mitlak BH. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. N Engl J Med. 2001 May 10;344(19):1434-41. doi: 10.1056/NEJM200105103441904. PMID 11346808
- [Background] Haas AV, LeBoff MS. Osteoanabolic Agents for Osteoporosis. J Endocr Soc. 2018 Jul 9;2(8):922-932. doi: 10.1210/js.2018-00118. eCollection 2018 Aug 1. PMID 30087947
- [Background] Lindsay R, Nieves J, Formica C, Henneman E, Woelfert L, Shen V, Dempster D, Cosman F. Randomised controlled study of effect of parathyroid hormone on vertebral-bone mass and fracture incidence among postmenopausal women on oestrogen with osteoporosis. Lancet. 1997 Aug 23;350(9077):550-5. doi: 10.1016/S0140-6736(97)02342-8. PMID 9284777
- [Background] Choi H, Magyar CE, Nervina JM, Tetradis S. Different duration of parathyroid hormone exposure distinctively regulates primary response genes Nurr1 and RANKL in osteoblasts. PLoS One. 2018 Dec 21;13(12):e0208514. doi: 10.1371/journal.pone.0208514. eCollection 2018. PMID 30576321
- [Background] Choudhary S, Santone E, Yee SP, Lorenzo J, Adams DJ, Goetjen A, McCarthy MB, Mazzocca AD, Pilbeam C. Continuous PTH in Male Mice Causes Bone Loss Because It Induces Serum Amyloid A. Endocrinology. 2018 Jul 1;159(7):2759-2776. doi: 10.1210/en.2018-00265. PMID 29757436
- [Background] Saag KG, Petersen J, Brandi ML, Karaplis AC, Lorentzon M, Thomas T, Maddox J, Fan M, Meisner PD, Grauer A. Romosozumab or Alendronate for Fracture Prevention in Women with Osteoporosis. N Engl J Med. 2017 Oct 12;377(15):1417-1427. doi: 10.1056/NEJMoa1708322. Epub 2017 Sep 11. PMID 28892457